CLINICAL TRIAL: NCT03590873
Title: The Effect of Restrictive Fluid and Vasopressin During Surgery of Burn Patients: a Randomized Clinical Trial
Brief Title: The Effect of Restrictive Fluid and Vasopressin During Surgery of Burn Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hee Yeong Kim, Assistant Professor, Hangang Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-051
Record Dates: First submitted 2018-06-28; First posted 2018-07-18 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Burn Surgery
MeSH Terms: interventions — Vasopressins; Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Intraoperative fluid management: administration of 6-10 ml/kg/hr of crystalloid solution.
- Restrictive group (Experimental): Intervention: administration of vasopressin 0.01 - 0.04 U/min after induction of anesthesia.
  Intraoperative fluid management: administration of 2-4 ml/kg/hr of crystalloid solution.
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — Vasopressin, is a hormone synthesized as a peptide prohormone in neurons in the hypothalamus, and is converted to arginine vasopressin. It then travels down the axon of that cell, which terminates in the posterior pituitary, and is released from vesicles into the circulation in response to extracellular fluid hypertonicity (hyperosmolality). Arginine vasopressin has two primary functions. First, it increases the amount of solute-free water reabsorbed back into the circulation from the filtrate in the kidney tubules of the nephrons. Second, arginine vasopressin constricts arterioles, which increases peripheral vascular resistance and raises arterial blood pressure.
  Other Names: Antidiuretic hormone, arginine vasopressin, or argipressin
  Arms: Restrictive group

SUMMARY:
This is a randomized double-blinded study to investigate in which the groups are designated as the control group and the restrictive group to further evaluate significant differences in intraoperative blood loos during burn surgery.

DETAILED DESCRIPTION:
This is a randomized double-blinded study to investigate the effect of fluid restriction and vasopressin on blood loss during surgery of the burn patients. The groups are designated as the control group and the restrictive group to further evaluate significant differences in intraoperative blood loss during the surgery.

ELIGIBILITY:
Inclusion criteria:

* age ≥ 18 years old
* burn patients undergoing surgery (TBSA > 20%)

Exclusion criteria:

* age < 18 years old
* history of renal disorder
* history of cardiac disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-06-04 (Estimated); Study Completion 2019-06-04 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | At the end of the surgery, approximately 3 hrs
  Comparison of the amounts of estimated blood loss in the two groups.

SECONDARY OUTCOMES:
Intraoperative red blood cell transfusion | At the end of the surgery, approximately 3 hrs
  Comparison of total units of red blood cell transfusion in the two groups.
Postoperative pulmonary complication | Within 7 postoperative days
  Comparison of postoperative pulmonary complication in the two groups.
Postoperative cardiovascular complication | Within 7 postoperative days
  Comparison of postoperative cardiovascular complication in the two groups.
Postoperative renal complication | Within 7 postoperative days
  Comparison of postoperative acute kidney injury in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, South Korea